CLINICAL TRIAL: NCT01632605
Title: Rapamycin in Advanced Polycystic Kidney Disease Pilot Study
Brief Title: The Vienna RAP Pilot Study
Acronym: RAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gere Sunder-Plassmann, Associate Professor of Medicine, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 003/2008/1.0
Record Dates: First submitted 2012-05-13; First posted 2012-07-03 (Estimated); Last update posted 2012-07-03 (Estimated); Status verified 2012-06

CONDITIONS: ADPKD
Keywords: ADPKD; Autosomal dominant polycystic kidney disease; Sirolimus; Rapamune; Polycystic liver disease; Rapamycin; Mammalian target of rapamycin; m-TOR; m-TOR inhibition
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Polycystic liver disease; Hereditary Sensory and Autonomic Neuropathies | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sirolimus (Experimental): Daily single oral dose of 1-3mg sirolimus with an initial loading dose of 6mg.
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Coated tablets, 1mg and 2mg available. Daily oral single dose with trough levels of 4-8ng/mL. Total intake for 6 months.
  Other Names: RAPAMUNE

SUMMARY:
The purpose of this study is to evaluate the safety of a daily single oral dose of sirolimus in patients with advanced autosomal dominant polycystic kidney disease.

DETAILED DESCRIPTION:
Autosomal dominant polycystic kidney disease (ADPKD) is the most common form of renal cystic diseases, affecting all ethnic groups with an incidence of 1 in 400 to 1.000. In Austria an estimated 8.000 to 21.000 people, and an estimated 670.000 to 1.675.000 people worldwide are affected by ADPKD, although statements of up to 6.000.000 affected individuals have been made. ADPKD is responsible for 5 to 10 percent of patients on chronic hemodialysis. Individuals with ADPKD usually present in the 3rd to 4th decade of life, progressing to end-stage renal disease within 5 to 10 years after the onset of renal insufficiency. Usually renal replacement therapy, either by chronic dialysis or renal transplantation, becomes necessary. Currently there is no treatment for ADPKD other than blood pressure control and supportive care.

Thus, novel therapies for ADPKD are of great importance.

The formation of cysts in ADPKD follows a mutation located within either the polycystic kidney disease 1 or -2 gene on chromosomes 16 and 4, which are coding for polycystin 1 (PC1) and -2 (PC2), respectively. PC1 and PC2 are members of the polycystin family of integral membrane proteins. PC1 acts as a G-protein coupled receptor and is suggested to mediate cell-cell and cell-matrix interactions. PC2 acts as a nonselective cation channel and is supposed to act in ion exchange mechanisms. Among other pathways PC1 and 2 are functioning via a mammalian target of rapamycin (mTOR) pathway, which is essential in protein translation, cell proliferation and -growth. Inhibition of the mTOR-pathway has reduced kidney enlargement in rodent polycystic kidney disease models and has shown to reduce the volume of cysts in human polycystic kidney- and polycystic liver disease. Thus, we hypothesize that the mTOR inhibitor sirolimus, an immunosuppressant drug with strong anti-proliferative effects, will delay the progression of renal insufficiency in patients with ADPKD in advanced stages of the disease.

Before conducting a large multicenter randomized controlled trial in this population we will demonstrate that therapy with mTOR-I does not accelerate the decline in renal function (as natural course of the disease), as well as mTOR-I does not aggravate prevalent-, or cause new onset of proteinuria, as expressed by the protein/creatinine ratio, in patients with ADPKD and an eGFR between 20 and 40 mL/min per 1.73sqm, compared to a historic cohort of patients with ADPKD and an eGFR between 20 and 40 mL/min per 1.73sqm, treated at the Department of Medicine III, Division of Nephrology and Dialysis, Medical University Vienna.

ELIGIBILITY:
Inclusion Criteria:

* ADPKD
* Eighteen years of age, or older.
* Baseline eGFR of 20-40mL/min per 1.73m2.
* Negative serum pregnancy test prior to administration of sirolimus and agreement to use contraception throughout the pilot safety study and three months after. Any participant who is getting pregnant during the pilot safety study period will have to discontinue.
* Written informed consent.

Exclusion Criteria:

* Pregnancy or lactation or plans to become pregnant in the near future or disagreement to use contraception.
* History of life threatening complications of ADPKD.
* Evidence of active systemic- or localized major infection.
* Evidence of infiltrate, cavities or consolidation on chest X-ray.
* Use of any investigational drug or -treatment up to 4 weeks prior to the enrolment and during the pilot safety study.
* Known hypersensitivity to sirolimus and its derivatives.
* Treatment with substances known to interfere with the cytochrome p-450 (CYP) 3A4/3A5 systems.
* Screening/baseline total white blood cell count below or equal to 3000/mm3.
* Screening/baseline platelet count below or equal to 100.000/mm3.
* Screening/baseline fasting triglycerides above or equal to 400 mg/dL.
* Screening/baseline fasting total cholesterol above or equal to 300 mg/dL.
* Concomitant glomerular diseases.
* Psychiatric disorders or any condition that might prevent the full comprehension of the purposes and risks of the pilot safety study.
* History of malignancies with the exception of adequately treated basal- and squamous-cell carcinomas of the skin.
* HIV infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-11; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Slope in estimated glomerular filtration rate (eGFR; 4 variables MDRD equation) and proteinuria within six months of exposure to sirolimus. | Six months
  A single daily oral dose of sirolimus with trough levels of 4 to 8ng/dL in patients with advanced polycystic kidney disease and an eGFR of 20-40mL/min per 1.73m2 does not lead to a greater decline in kidney function as represented by the eGFR than -8.8mL/min per 1.73m2 within 6 months (one-sided) as well as it does not lead to an incline in proteinuria, as represented by the logarithm of the protein-creatinine ratio, greater than 0.39 within 6 months (one-sided).

SECONDARY OUTCOMES:
Leucopenia | 6 months
  Drop in WBC below 4 G/L
Thrombopenia | 6 months
  Drop in platelets below 150 G/L
Aphthae | 6 months
  New onset of aphthaeous stomatitis under therapy with sirolimus
Dysfunctional wound healing | 6 months
  Dysfunctional and/or prolonged wound healing attributed to sirolimus therapy
Pneumonitis | 6 months
  Persisting cough and infiltrates on chest x-ray
Acne | 6 months
  Acne attributed to sirolimus therapy

CONTACTS AND LOCATIONS:
Overall Officials: Gere Sunder-Plassmann, MD, Principal Investigator — Medical University Vienna
Locations (1):
- Division of Nephrology and Dialysis, Department of Medicine III, Medical University Vienna, Vienna, Vienna, Austria